CLINICAL TRIAL: NCT02548663
Title: Sport Therapy for Contrasting the Deterioration of Muscle Oxidative Metabolism in Patients Affected by Amyotrophic Lateral Sclerosis (ALS) - Project ME_E_SLA
Brief Title: Sport Therapy and Osteopathy Manipulative Treatment in ALS
Acronym: ME_E_SLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: Italian Academy of Osteopathic Medicine (AIMO), Saronno, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ME_E_SLA
Record Dates: First submitted 2015-09-02; First posted 2015-09-14 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; sport therapy; osteopathic manual treatment; muscle oxidative metabolism
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active; sport therapy (Experimental): active exercise carefully calibrated on residual capacities.
  Interventions: Other: Sport therapy
- passive; osteopathic treatment (Experimental): manipulative treatment according to osteopathic principles.
  Interventions: Other: Osteopathic treatment

INTERVENTIONS:
Other: Sport therapy — Frequency: 60 min three times/week
  1. 20 min: aerobic training on bicycle ergometer.
  2. 20 min: strength training at 60% of maximal load.
  3. 20 min: proprioception and stretching exercises.
  Arms: active; sport therapy
Other: Osteopathic treatment — Frequency: 60 min weekly
  Arms: passive; osteopathic treatment

SUMMARY:
This project assessed muscle oxidative metabolism and fatigue in patients affected by amyotrophic lateral sclerosis (ALS) undergoing to three months of individualized cardiovascular and strength training. Muscle oxidative metabolism and strength will be assessed by non-invasive methods, such as near-infrared spectroscopy (NIRS) and mechanomyography (MMG). NIRS is a technique giving indications on the capacity of oxygen extraction of muscles during exercise. MMG allows analyzing the pattern of motor unit recruitment and related fatigue. The investigators will also assess the effects of training on pain tolerance and quality of life (QoL) by the Brief Pain Inventory and the McGill Quality of Life questionnaires, using the validated Italian versions. Patients will be assessed longitudinally before (time T0) and after three months of individualized training (time T1). After one month of de-training (time T2) the investigators will assess the hypothetic persistence of any treatment-related effect. The effect of three months-osteopathic treatment (osteo) on pain and QoL will be assessed as well.

DETAILED DESCRIPTION:
Single blind pilot trial assessing the efficacy and side effects of active training or osteopathic manipulative treatment in ALS.

Interventions will be administered for three months (plus one month without intervention) by specialized personnel.

Primary outcome measures will include: exercise tolerance and muscle oxygen extraction capacity, side effects. Secondary outcome measures will include: pain, QoL and disease progression scales.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ALS
* early stages of disease
* able to perform exercise with major muscle groups.

Exclusion Criteria:

* non-invasive ventilation (NIV)
* tracheostomy
* coronaropathy
* ongoing infectious diseases
* cognitive deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
change in the relationship between maximal oxygen consumption (VO2max) and muscle oxygen extraction capacity at 12 weeks | 12 weeks
  exercise tolerance assessed by Cardio pulmonary Exercise Test (CPET); oxygen extraction on vastus lateralis, respiratory muscle and hand thenar eminence muscles assessed by Near Infrared Spectroscopy (NIRS)
appearance of side effects during the period of intervention administration | 12 weeks

SECONDARY OUTCOMES:
change of pain at 12 weeks | 12 weeks
  Brief Pain Inventory (BPI)
change of quality of life at 12 weeks | 12 weeks
  McGill Quality of Life
change of the neurological functional status at 12 weeks | 12 weeks
  ALS Functional Rating Scale-revised (ALSFRS-R)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Lanfranconi, MD, Principal Investigator — University of Milano Bicocca

REFERENCES:
- [Background] Arbesman M, Sheard K. Systematic review of the effectiveness of occupational therapy-related interventions for people with amyotrophic lateral sclerosis. Am J Occup Ther. 2014 Jan-Feb;68(1):20-6. doi: 10.5014/ajot.2014.008649. PMID 24367951
- [Background] Bohannon RW. Results of resistance exercise on a patient with amyotrophic lateral sclerosis. A case report. Phys Ther. 1983 Jun;63(6):965-8. doi: 10.1093/ptj/63.6.965. PMID 6856684
- [Background] Caraceni A, Mendoza TR, Mencaglia E, Baratella C, Edwards K, Forjaz MJ, Martini C, Serlin RC, de Conno F, Cleeland CS. A validation study of an Italian version of the Brief Pain Inventory (Breve Questionario per la Valutazione del Dolore). Pain. 1996 Apr;65(1):87-92. doi: 10.1016/0304-3959(95)00156-5. PMID 8826494
- [Background] Carilho R, de Carvalho M, Swash M, Pinto S, Pinto A, Costa J. Vascular endothelial growth factor and amyotrophic lateral sclerosis: the interplay with exercise and noninvasive ventilation. Muscle Nerve. 2014 Apr;49(4):545-50. doi: 10.1002/mus.23955. PMID 23868282
- [Background] Carreras I, Yuruker S, Aytan N, Hossain L, Choi JK, Jenkins BG, Kowall NW, Dedeoglu A. Moderate exercise delays the motor performance decline in a transgenic model of ALS. Brain Res. 2010 Feb 8;1313:192-201. doi: 10.1016/j.brainres.2009.11.051. Epub 2009 Dec 5. PMID 19968977
- [Background] Chio A, Canosa A, Gallo S, Moglia C, Ilardi A, Cammarosano S, Papurello D, Calvo A. Pain in amyotrophic lateral sclerosis: a population-based controlled study. Eur J Neurol. 2012 Apr;19(4):551-5. doi: 10.1111/j.1468-1331.2011.03540.x. Epub 2011 Oct 4. PMID 21972798
- [Background] Colombo R, Mazzini L, Mora G, Parenzan R, Creola G, Pirali I, Minuco G. Measurement of isometric muscle strength: a reproducibility study of maximal voluntary contraction in normal subjects and amyotrophic lateral sclerosis patients. Med Eng Phys. 2000 Apr;22(3):167-74. doi: 10.1016/s1350-4533(00)00024-2. PMID 10964037
- [Background] Dal Bello-Haas V, Florence JM. Therapeutic exercise for people with amyotrophic lateral sclerosis or motor neuron disease. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD005229. doi: 10.1002/14651858.CD005229.pub3. PMID 23728653
- [Background] Bello-Haas VD, Florence JM, Kloos AD, Scheirbecker J, Lopate G, Hayes SM, Pioro EP, Mitsumoto H. A randomized controlled trial of resistance exercise in individuals with ALS. Neurology. 2007 Jun 5;68(23):2003-7. doi: 10.1212/01.wnl.0000264418.92308.a4. PMID 17548549
- [Background] Deforges S, Branchu J, Biondi O, Grondard C, Pariset C, Lecolle S, Lopes P, Vidal PP, Chanoine C, Charbonnier F. Motoneuron survival is promoted by specific exercise in a mouse model of amyotrophic lateral sclerosis. J Physiol. 2009 Jul 15;587(Pt 14):3561-72. doi: 10.1113/jphysiol.2009.169748. Epub 2009 Jun 2. PMID 19491245
- [Background] Drory VE, Goltsman E, Reznik JG, Mosek A, Korczyn AD. The value of muscle exercise in patients with amyotrophic lateral sclerosis. J Neurol Sci. 2001 Oct 15;191(1-2):133-7. doi: 10.1016/s0022-510x(01)00610-4. PMID 11677004
- [Background] Kirkinezos IG, Hernandez D, Bradley WG, Moraes CT. Regular exercise is beneficial to a mouse model of amyotrophic lateral sclerosis. Ann Neurol. 2003 Jun;53(6):804-7. doi: 10.1002/ana.10597. PMID 12783429
- [Background] Mahoney DJ, Rodriguez C, Devries M, Yasuda N, Tarnopolsky MA. Effects of high-intensity endurance exercise training in the G93A mouse model of amyotrophic lateral sclerosis. Muscle Nerve. 2004 May;29(5):656-62. doi: 10.1002/mus.20004. PMID 15116368
- [Background] Pinto AC, Alves M, Nogueira A, Evangelista T, Carvalho J, Coelho A, de Carvalho M, Sales-Luis ML. Can amyotrophic lateral sclerosis patients with respiratory insufficiency exercise? J Neurol Sci. 1999 Oct 31;169(1-2):69-75. doi: 10.1016/s0022-510x(99)00218-x. PMID 10540010
- [Background] Veldink JH, Bar PR, Joosten EA, Otten M, Wokke JH, van den Berg LH. Sexual differences in onset of disease and response to exercise in a transgenic model of ALS. Neuromuscul Disord. 2003 Nov;13(9):737-43. doi: 10.1016/s0960-8966(03)00104-4. PMID 14561497